CLINICAL TRIAL: NCT05497648
Title: Choose to Move: Impact and Implementation Evaluation of a Program to Enhance Older Adult Physical Activity, Mobility and Health
Brief Title: Evaluating Impact and Implementation of Choose to Move (Phase 3)
Acronym: CTM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Active Aging Society (Other)
Responsible Party: Principal Investigator, Heather McKay, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H15-02522; PJT-153248 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2022-08-05; First posted 2022-08-11 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Aging; Physical Inactivity; Mobility Limitation; Loneliness; Social Isolation
Keywords: implementation science; scale-up; behaviour change; physical activity; mobility; loneliness; social connectedness; social isolation; older adults; fidelity; adaptation
MeSH Terms: conditions — Sedentary Behavior; Mobility Limitation; Social Isolation; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Choose to Move (Experimental): Individuals responsible for delivering Choose to Move and older adults enrolled in Choose to Move
  Interventions: Behavioral: Choose to Move

INTERVENTIONS:
Behavioral: Choose to Move — CTM (phase 3) is a 6-month, flexible, evidence- and choice-based program for low active older adults.
  CTM includes
  * One-on-One Consultation Participants meet 1-on-1 with their activity coach at the start of the program to set goals and develop an action plan tailored to their abilities, interests and resources. Older adults can choose to participate in individual or group-based activities.
  * Group Meetings Over the first three months, participants will attend five, 1-hour group-based meetings (up to 12 participants total) led by their activity coach. Meetings cover a discussion topic and provide time and space for social connection between participants.
  * Check-ins Over the six month program, activity coaches will provide six brief telephone check-ins (approximately 15 minutes each and once/month) to discuss their Action Plan and ask questions.
  Other Names: CTM

SUMMARY:
The objectives of this study are to 1) evaluate whether Choose to Move (CTM) improves health outcomes in older adults who participate and 2) assess whether CTM is delivered as planned and what factors support or inhibit delivery at scale.

CTM is a 6 month, choice-based program for low active older adults being scaled-up across British Columbia, Canada. The goals of CTM are to enhance physical activity, mobility and social connectedness in older adults living in British Columbia, Canada.

DETAILED DESCRIPTION:
CTM is a 6 month, choice-based program for low active older adults being scaled-up in phases across British Columbia, Canada. Within CTM (phase 3), trained activity coaches support older adults in three ways. First, in a one-on-one consultation, activity coaches help participants to set goals and create action plans for physical activity tailored to each person's interests and abilities. Older adults can choose to participate in individual or group-based activities. Second, activity coaches facilitate a series of group meetings with small groups of participants. Finally, activity coaches regularly check in with participants to provide ongoing support. Activity coaches and recreation departments across BC are trained and provided with resources to deliver CTM.

Objectives:

1. To assess the impact (effectiveness) of CTM (phase 3) delivered at scale on the physical activity, mobility and social connectedness of older adults (Part I - Impact Evaluation)
2. To assess whether the program was implemented as planned (fidelity) and investigate factors that support or inhibit implementation at scale (Part II - Implementation Evaluation).

Study Design:

We use a hybrid type 2 effectiveness-implementation (Curran et al 2012) pre-post study design to evaluate CTM. We use mixed-methods (quantitative and qualitative) and collect data at 0 (baseline), 3 (mid-intervention), 6 (post-intervention) and 18 (12-months post-intervention) months to assess effectiveness and implementation of CTM.

ELIGIBILITY:
Inclusion Criteria (older adults):

* ≥60 years of age,
* demonstrate readiness for physical activity via the PAR-Q+ questionnaire (Warburton et al 2011), Get Active Questionnaire (Canadian Society for Exercise Physiology 2017) or a letter of recommendation from their physician
* <150 min/week physical activity
* English speaking

Exclusion Criteria (older adults):

- previous participation in CTM

Inclusion Criteria (delivery partners):

* Activity coaches will be English speaking BCRPA Registered Older Adult Fitness Leaders or Kinesiologists who are delivering CTM at participating centres
* Recreation Managers and Coordinators affiliated with participating centres delivering CTM
* Provincial Partners (e.g., individuals/partners who make strategic and/or policy decisions) at partner organizations delivering Choose to Move

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1216 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Change in physical activity | 0, 3, 6, 18-months
  The single item physical activity questionnaire will be used to measure physical activity (Milton, Bull & Bauman, 2011). Output variable is self-reported number of days/week ≥30 min PA in the past week.

SECONDARY OUTCOMES:
Change in loneliness | 0, 3, 6, 18-months
  The three-item loneliness scale (Hughes et al., 2004) will be used to assess change in loneliness. Participants rate three aspects of loneliness. The output variable is loneliness score (range 3-9); lower scores indicate lower levels of loneliness.
Change in social isolation | 0, 3, 6, 18-months
  We assessed social isolation using a three-item questionnaire adapted from two questions on social contact frequency (Veroff et al 1981). The output variable is social isolation score (range 0-15); higher scores indicate less social isolation.
Change in physical functioning | 0, 3, 6, 18-months
  Mobility will be assessed with the Physical Functioning Subscale of the 36-Item Short Form Survey (SF-36; Ware et al., 1989). The measure asks participants to rate if their health limits them in performing 10 different activities. The output variable is an average score from 0-100 of physical functioning, where a higher score indicates a more favourable health state.
Change in physical activity (PAAQ) | 0, 3, 6, 18-months
  The Physical Activity Adult Questionnaire will be used to assess physical activity over the previous 7 days (Garriguet et al 2015). Output variable is minutes of PA/week.
Change in health-related quality of life (EQ-5D-5L Profile) | 0, 3, 6, 18-months
  Health status (EQ-5D-5L Profile) will be assessed with the EQ-5D-5L (The EuroQol Group, 1990). Participants report on mobility, self-care, usual activities, pain/discomfort and anxiety/depression on a scale from 1-5 (level of perceived problems) for each item. Responses are used to create a 5-digit number which will be used descriptively.
Change in health-related quality of life (EQ-5D-5L Level Sum Score) | 0, 3, 6, 18-months
  Health status (EQ-5D-5L Level Sum Score) will be assessed with the EQ-5D-5L (The EuroQol Group, 1990). Participants report on mobility, self-care, usual activities, pain/discomfort and anxiety/depression on a scale from 1-5 (level of perceived problems) for each item. The Level Sum Score uses the 5-digit profile to create a numeric score, with scores ranging from 5-25 (lower levels indicate lower levels of perceived problems).
Change in health-related quality of life (EQ-5D-5L Visual Analogue Scale) | 0, 3, 6, 18-months
  health status (EQ-5D-5L Visual Analogue Scale) will be assessed with the EQ-5D-5L (The EuroQol Group, 1990). Participants report on their health on a visual analogue scale from 0 (worst health) to 100 (best health).
Change in mobility limitations | 0, 3, 6, 18-months
  Two items will assess change in a participants' ability to walk a quarter of a mile and up 10 steps (Simonsick et al., 2008). The output variable is self-reported presence of mobility-disability (no/any difficulty walking 400m or climbing one flight of stairs).
Change In sitting time | 0, 3, 6, 18-months
  A five-item questionnaire (Marshall et al., 2010) will be used to assess change in sitting time (hours and minutes) each day in the following domains: (a) while travelling to and from places (e.g., work, shops); (b) while at work; (c) while watching television; (d) while using a computer at home; and (e) at leisure not including watching television (e.g., visiting friends, movies, eating out) on a weekday and a weekend day. The output variables are sitting hours per day across 5 domains
Change in social network | 0, 3, 6, 18-months
  We use a six-item questionnaire (Lubben et al., 2006) to assess social isolation. The output variable is an equally weighted sum (range 0-30).
Change in grip strength (subset) | 0, 3, 6, 18-months
  We assess grip strength using a hand grip dynamometer and standard protocols. We combine the best trial from each side and report the sum as total grip strength.
Change in lower extremity function (subset) | 0, 3, 6, 18-months
  We use the short performance physical battery (SPPB) to assess lower extremity functioning (Guralnik et al 1994). The output variable is an equally weighted sum of 3 subscores (range 0-12); higher scores represent better performance.
Change in physical activity (CHAMPS) | 0, 3, 6, 18-months
  We use the CHAMPS questionnaire (Stewart et al 2001) to assess weekly frequency and duration of a variety of physical activities and use the CHAMPS scoring algorithms to calculate energy expenditure (kcal/week) and frequency (times/week).

OTHER OUTCOMES:
Reach-individual | 6 months
  The number of participants engaged in the intervention is obtained from program records.
Reach-organizational | 6 months
  The number of organizations and activity coaches delivering the intervention is obtained from program records.
Dose | 6 months
  The amount of intervention delivered is assessed via survey (designed in house)
Fidelity | 6 months
  Fidelity to planned delivery is assessed via survey (designed in house) and interview/focus group.
Participant responsiveness | 6 months
  We assess program satisfaction via participant survey (designed in house) and interviews.
Adaptation | 6 months
  We assess adaptation of the intervention and its delivery via survey (designed in house) and interview/focus groups
Contextual factors influencing implementation | 6 months
  We use surveys (designed in house) and interviews/focus groups to describe how community level factors, provider characteristics, characteristics of the innovation, the prevention delivery system, organizational capacity and the prevention support system influenced program delivery.
Cost | 6 months
  We use a cost capture template to record program delivery costs.

CONTACTS AND LOCATIONS:
Overall Officials: Heather A McKay, Principal Investigator — University of British Columbia; Joanie Sims Gould, Principal Investigator — University of British Columbia; Matthew Herman, MSc, Principal Investigator — Ministry of Health, British Columbia; Adrian Bauman, PhD, Principal Investigator — University of Sydney; Dawn Mackey, PhD, Principal Investigator — Simon Fraser University; Karim Miran-Khan, PhD, Principal Investigator — University of British Columbia; Patti-Jean Naylor, PhD, Principal Investigator — University of Victoria; Paul Stolee, PhD, Principal Investigator — University of Waterloo
Locations (1):
- Centre for Hip Health and Mobility, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Canadian Society for Exercise Physiology. Get Active Questionnaire. 2017. Available: https://csep.ca/wp-content/uploads/2021/05/GETACTIVEQUESTIONNAIRE_ENG.pdf
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Durlak JA, DuPre EP. Implementation matters: a review of research on the influence of implementation on program outcomes and the factors affecting implementation. Am J Community Psychol. 2008 Jun;41(3-4):327-50. doi: 10.1007/s10464-008-9165-0. PMID 18322790
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Garriguet D, Tremblay S, Colley RC. Comparison of Physical Activity Adult Questionnaire results with accelerometer data. Health Rep. 2015 Jul;26(7):11-7. PMID 26177042
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Lubben J, Blozik E, Gillmann G, Iliffe S, von Renteln Kruse W, Beck JC, Stuck AE. Performance of an abbreviated version of the Lubben Social Network Scale among three European community-dwelling older adult populations. Gerontologist. 2006 Aug;46(4):503-13. doi: 10.1093/geront/46.4.503. PMID 16921004
- [Background] Marshall AL, Miller YD, Burton NW, Brown WJ. Measuring total and domain-specific sitting: a study of reliability and validity. Med Sci Sports Exerc. 2010 Jun;42(6):1094-102. doi: 10.1249/MSS.0b013e3181c5ec18. PMID 19997030
- [Background] Milton K, Bull FC, Bauman A. Reliability and validity testing of a single-item physical activity measure. Br J Sports Med. 2011 Mar;45(3):203-8. doi: 10.1136/bjsm.2009.068395. Epub 2010 May 19. PMID 20484314
- [Background] Milton K, Clemes S, Bull F. Can a single question provide an accurate measure of physical activity? Br J Sports Med. 2013 Jan;47(1):44-8. doi: 10.1136/bjsports-2011-090899. Epub 2012 Apr 20. PMID 22522584
- [Background] Simonsick EM, Newman AB, Visser M, Goodpaster B, Kritchevsky SB, Rubin S, Nevitt MC, Harris TB; Health, Aging and Body Composition Study. Mobility limitation in self-described well-functioning older adults: importance of endurance walk testing. J Gerontol A Biol Sci Med Sci. 2008 Aug;63(8):841-7. doi: 10.1093/gerona/63.8.841. PMID 18772472
- [Background] Stewart AL, Mills KM, King AC, Haskell WL, Gillis D, Ritter PL. CHAMPS physical activity questionnaire for older adults: outcomes for interventions. Med Sci Sports Exerc. 2001 Jul;33(7):1126-41. doi: 10.1097/00005768-200107000-00010. PMID 11445760
- [Background] Veroff, J.; Kulka, R. A.; Douvan, E. Mental health in America: Patterns of help-seeking from 1957-1976. Basic Books: New York, 1981.
- [Background] Warburton DE, Jamnik VK, Bredin SSD, Gledhill N, on behalf of the PAR-Q+ Collaboration. The Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) and Electronic Physical Activity Readiness Medical Examination (ePARmed-X+). Health & Fitness Journal of Canada. 2011;4(2):3-23.
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- See also: Website for the Choose to Move Program — https://www.choosetomove.ca/